CLINICAL TRIAL: NCT00777036
Title: A Phase II Study of Dasatinib Therapy in Children and Adolescents With Newly Diagnosed Chronic Phase Chronic Myelogenous Leukemia or With Ph+ Leukemias Resistant or Intolerant to Imatinib
Brief Title: A Phase II Study of Dasatinib in Children and Adolescents With Newly Diagnosed Chronic Phase Chronic Myelogenous Leukemia (CML) or With Ph+ Leukemias Resistant or Intolerant to Imatinib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA180-226; 2008-002260-33 (EudraCT Number)
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Results first posted 2018-01-05 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Leukemia
Keywords: Leukemia, Pediatric
MeSH Terms: conditions — Leukemia | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: Imatinib-resistant/intolerant CP-CML (Experimental): Dasatinib 60 mg/m² tablet every day (QD) [with a maximum dose of 100 mg QD for subjects with high BSA] for minimum of 24 months, may continue as long as deriving clinical benefit
  OR
  Dasatinib 72 mg/m² powder for oral suspension (PFOS) QD [with a maximum dose of 120 mg QD for subjects with high BSA] for minimum of 24 months, may continue as long as deriving clinical benefit
  Interventions: Drug: Dasatinib
- Cohort 2: Ph+ALL or AP- or BP-CML (Experimental): Dasatinib 80 mg/m² tablet QD [with a maximum dose of 140 mg QD for subjects with high BSA] for minimum of 24 months, may continue as long as deriving clinical benefit
  OR
  Dasatinib 96 mg/m² PFOS QD [with a maximum dose of 170 mg QD for subjects with high BSA] for minimum of 24 months, may continue as long as deriving clinical benefit
  Interventions: Drug: Dasatinib
- Cohort 3: Newly diagnosed, treatment naïve CP-CML (Experimental): Dasatinib 60 mg/m² tablet QD [with a maximum dose of 100 mg QD for subjects with high BSA] for minimum of 24 months, may continue as long as deriving clinical benefit
  OR
  Dasatinib 72 mg/m² PFOS QD [with a maximum dose of 120 mg QD for subjects with high BSA] for minimum of 24 months, may continue as long as deriving clinical benefit
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib
  Other Names: Sprycel (BMS-354825)

SUMMARY:
The purpose of this study is to determine whether dasatinib is safe and effective in children and adolescents with newly diagnosed chronic myeloid leukemia (CML), or in children with Ph+ acute lymphoblastic leukemia (ALL), accelerated or blast phases CML who relapse after imatinib or who are resistant or intolerant to imatinib. The side effects of this oral investigational drug in children and adolescents will be evaluated

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* CP-CML who prove resistant or intolerant to imatinib (Cohort 1)
* Ph+ ALL, AP-CML, or BP-CML who are resistant or intolerant to or who relapse after imatinib therapy (Cohort 2)
* Newly diagnosed, treatment naive CP-CML (Cohort 3)
* Lansky or Karnofsky scale >50
* Life expectancy ≥12 weeks
* Adequate hepatic and renal function
* Written informed consent
* Target Population for the PK substudy must obtain written informed consent from subject, or from parents or legal guardians for minor subjects, according to local law and regulation
* Target Population for the PK substudy subjects must have CP-CML and be taking daily dasatinib (tablets or PFOS) either as part of Cohort 1 or Cohort 3 of this protocol. Patients receiving commercial dasatinib tablets outside of this protocol may be invited to participate in this PK substudy
* Target Population for the PK substudy subjects with CP-CML who are tolerating dasatinib tablet dose of at least 60 mg/m2 or dasatinib PFOS dose of at least 72 mg/m2
* Target Population for the PK substudy prior exposure to imatinib or other TKI therapy is permissible
* Target Population for the PK substudy subjects must meet relevant inclusion criteria

Exclusion Criteria:

* Eligibility for potentially-curative therapy including hematopoietic stem-cell transplantation
* Symptomatic CNS involvement (other than signs and symptoms caused by leptomeningeal disease)
* Isolated extramedullary disease
* Prior therapy with Dasatinib
* Target Population for the PK substudy subjects participating in the PK substudy must comply with the relevant exclusion criteria
* Target Population for the PK substudy subjects are not allowed to use proton pump inhibitors, H2 antagonists, CYP3A4 inhibitors and inducers when entering the PK substudy

Other inclusion/exclusion criteria may apply

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 133 (Actual)
Dates: Start 2009-03-20 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2025-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (162):
- United States (33):
  - Local Institution, Birmingham, Alabama
  - Local Institution - 0005, Phoenix, Arizona
  - Phoenix Children'S Hospital, Phoenix, Arizona
  - Jonathan Jaques Children'S Cancer Center, Long Beach, California
  - Local Institution - 0001, Long Beach, California
  - Children'S Hospital Of Orange County, Orange, California
  - Local Institution - 0024, Orange, California
  - Children'S Hospital, Aurora, Colorado
  - Local Institution - 0004, Aurora, Colorado
  - Children's Healthcare Of Atlanta - Egleston, Atlanta, Georgia
  - Local Institution - 047, Atlanta, Georgia
  - Children's Hospital of Chicago, Chicago, Illinois
  - Local Institution - 0072, Chicago, Illinois
  - Local Institution, Chicago, Illinois
  - Dana Faber Cancer Institute, Boston, Massachusetts
  - Dana Farber Cancer Institute., Boston, Massachusetts
  - Local Institution - 0040, Boston, Massachusetts
  - Stephen D. Hassenfeld Children'S Center, New York, New York
  - Local Institution - 0061, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, New York, New York
  - Oregon Health & Sci Univ, Portland, Oregon
  - Local Institution - 0002, Portland, Oregon
  - Children'S Hospital Of Philadelphia, Philadelphia, Pennsylvania
  - Local Institution - 0014, Philadelphia, Pennsylvania
  - Children'S Hospital Of Pittsburgh, Pittsburgh, Pennsylvania
  - Local Institution - 0003, Pittsburgh, Pennsylvania
  - Local Institution - 0035, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Local Institution - 0048, Houston, Texas
  - Texas Children'S Cancer Center, Houston, Texas
  - Local Institution - 0028, Seattle, Washington
  - Seattle Children'S, Seattle, Washington
- Argentina (6):
  - Local Institution - 0043, Bunos Aires, Buenos Aires
  - Local Institution, Bunos Aires, Buenos Aires
  - Hospital Nacional Profesor Alejandro Posadas, El Palomar, Buenos Aires
  - Local Institution - 0049, El Palomar, Buenos Aires
  - Local Institution - 0042, Córdoba
  - Local Institution, Córdoba
- Australia (10):
  - Local Institution - 065, Randwick, New South Wales
  - Local Institution, Randwick, New South Wales
  - Local Institution - 069, Westmead, New South Wales
  - Local Institution, Westmead, New South Wales
  - Local Institution - 0064, Sth Brisbane, Queensland
  - Local Institution, Sth Brisbane, Queensland
  - Local Institution - 067, North Adelaide, South Australia
  - Local Institution, North Adelaide, South Australia
  - Local Institution - 0066, Parkville, Victoria
  - Local Institution, Parkville, Victoria
- Brazil (9):
  - Local Institution - 0021, Curitiba, Paraná
  - Local Institution, Curitiba, Paraná
  - Local Institution - 0022, Porto Alegre, Rio Grande do Sul
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0019, São Paulo, São Paulo
  - Local Institution - 0020, Campinas
  - Local Institution, Campinas
  - Local Institution - 0039, São Paulo
  - Local Institution, São Paulo
- Canada (14):
  - Alberta Children'S Hospital, Calgary, Alberta
  - Local Institution - 0079, Calgary, Alberta
  - Local Institution - 0078, Edmonton, Alberta
  - Stollery Children'S Hospital, Edmonton, Alberta
  - Bc Children'S Hospital, Vancouver, British Columbia
  - Local Institution - 077, Vancouver, British Columbia
  - Iwk Health Centre, Halifax, Nova Scotia
  - Local Institution - 073, Halifax, Nova Scotia
  - Children'S Hospital Of Eastern Ontario, Ottawa, Ontario
  - Local Institution - 086, Ottawa, Ontario
  - Local Institution - 076, Toronto, Ontario
  - The Hospital For Sick Children, Toronto, Ontario
  - Chu Ste-Justine, Montreal, Quebec
  - Local Institution - 080, Montreal, Quebec
- France (9):
  - Local Institution - 0030, Lyon
  - Local Institution, Lyon
  - Local Institution - 0032, Nantes
  - Local Institution, Nantes
  - Local Institution - 0037, Paris
  - Local Institution, Paris
  - Local Institution - 0029, Paris
  - Local Institution - 036, Poitiers
  - Local Institution, Poitiers
- Germany (4):
  - Local Institution - 075, Frankfurt
  - Local Institution, Frankfurt
  - Local Institution - 0074, Hanover
  - Local Institution, Hanover
- India (16):
  - Local Institution - 0089, Navrangpura, Ahmedabad, Gujarat
  - Local Institution, Navrangpura, Ahmedabad, Gujarat
  - Local Institution, Bangalore, Karnataka
  - Local Institution, Mumbai, Maharashtra
  - Local Institution - 0094, Pune, Maharashtra
  - Local Institution, Pune, Maharashtra
  - Local Institution - 0093, Madurai, Tamil Nadu
  - Local Institution, Madurai, Tamil Nadu
  - Local Institution, Vellore, Tamil Nadu
  - Local Institution - 0088, Bangalore
  - Local Institution - 0082, Kolkata
  - Local Institution, Kolkata
  - Local Institution - 0085, Mumbai
  - Local Institution, Mumbai
  - Local Institution - 0084, Trivandrum
  - Local Institution, Trivandrum
- Italy (9):
  - Local Institution - 038, Bologna
  - Local Institution, Bologna
  - Local Institution - 006, Monza
  - Local Institution, Monza (MB)
  - Local Institution - 070, Roma
  - Local Institution, Roma
  - Local Institution - 0059, Roma
  - Local Institution - 015, Torino
  - Local Institution, Torino
- Mexico (12):
  - Hospital Civil De Guadalajara - Nuevo Dr. Juan I. Menchaca, Guadalajara, Jalisco
  - Local Institution - 0054, Guadalajara, Jalisco
  - Local Institution - 0051, Cuauhtémoc, Mexico City
  - Local Institution, Df, Mexico City
  - Local Institution - 0053, Mexico City, Mexico City
  - Local Institution, Mexico City, Mexico City
  - Local Institution - 0052, Mexico City, Mexico City
  - Local Institution, Mexico, D. F., Mexico City
  - Local Institution - 0050, Monterrey, Nuevo León
  - Local Institution, Monterrey, Nuevo León
  - Local Institution - 0060, Monterrey, N.l., Nuevo León
  - Local Institution, Monterrey, N.l., Nuevo León
- Netherlands (3):
  - Local Institution - 0007, Rotterdam
  - Local Institution, Rotterdam
  - Local Institution - 0099, Utrecht
- Romania (3):
  - Local Institution - 0095, Bucharest
  - Local Institution, Bucharest
  - Local Institution - 0097, Sector 2
- Russia (5):
  - Local Institution - 0017, Moscow
  - Local Institution, Moscow
  - Local Institution - 0023, Moscow
  - Local Institution - 0018, Saint Petersburg
  - Local Institution, Saint Petersburg
- Singapore (2):
  - Local Institution - 0071, Singapore
  - Local Institution, Singapore
- South Africa (8):
  - Local Institution - 0055, Bloemfontein, Free State
  - Local Institution, Bloemfontein, Free State
  - Local Institution - 058, Pretoria, Gauteng
  - Local Institution, Pretoria, Gauteng
  - Local Institution - 0057, Cape Town, Western Cape
  - Local Institution, Cape Town, Western Cape
  - Local Institution - 062, Tygerberg, Western Cape
  - Local Institution, Tygerberg, Western Cape
- South Korea (3):
  - Local Institution - 0092, Seoul
  - Local Institution, Seoul
  - Local Institution - 0091, Seoul
- Spain (10):
  - Local Institution - 0013, Barcelona
  - Local Institution, Barcelona
  - Local Institution - 0012, Barcelona
  - Local Institution - 0011, Madrid
  - Local Institution, Madrid
  - Local Institution - 0010, Madrid
  - Local Institution - 0041, Málaga
  - Local Institution, Málaga
  - Local Institution - 0033, Valencia
  - Local Institution, Valencia
- United Kingdom (6):
  - Local Institution - 0016, Glasgow, Central
  - Local Institution, Glasgow, Central
  - Local Institution - 0009, Sutton, Surrey
  - Local Institution, Sutton, Surrey
  - Local Institution - 0008, Birmingham, West Midlands
  - Local Institution, Birmingham, West Midlands

REFERENCES:
- [Derived] Gore L, Kearns PR, de Martino ML, Lee, De Souza CA, Bertrand Y, Hijiya N, Stork LC, Chung NG, Cardos RC, Saikia T, Fagioli F, Seo JJ, Landman-Parker J, Lancaster D, Place AE, Rabin KR, Sacchi M, Swanink R, Zwaan CM. Dasatinib in Pediatric Patients With Chronic Myeloid Leukemia in Chronic Phase: Results From a Phase II Trial. J Clin Oncol. 2018 May 1;36(13):1330-1338. doi: 10.1200/JCO.2017.75.9597. Epub 2018 Mar 2. PMID 29498925
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 80 sites (Argentina, Australia, Brazil, Canada, France, Germany, Great Britain, India, Italy, Korea, Mexico, Netherlands, Romania, Russia, Singapore, South Africa, Spain, and USA).
Pre-assignment Details: The PK sub-study analysis is not part of the pre-specified primary and secondary outcome measures.
Groups:
- Cohort 1: Children and adolescents with CP-CML who were resistant or intolerant to imatinib received dasatinib tablets at 60 mg/m2 QD on a continuous oral regimen.
- Cohort 2: Children and adolescents with Ph+ ALL, AP-CML or BP-CML who were resistant or intolerant to, or relapsed after imatinib therapy received dasatinib tablets at a dose schedule of 80 mg/m2 QD on a continuous oral regimen.
- Cohort 3: Children and adolescents with CP-CML who were treatment-naive received dasatinib tablets at 60 mg/m2 QD or powder for oral suspension (PFOS) at 72 mg/m2 QD on a continuous oral regimen.
- PK Sub-Study: Children and adolescents received powder for oral suspension (PFOS) at a dose of 90 mg/m2 QD to evaluate the pharmacokinetics of dasatinib.
Period: On Treatment
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | PK Sub-Study
Started | 29 | 17 | 84 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 29 | 17 | 84 | 0
Not completed — Reached 18 years of age and transitioned to commercial drug | 13 | 7 | 42 | 0
Not completed — Administrative Reason By Sponsor | 1 | 0 | 9 | 0
Not completed — Failure to Meet Study Criteria | 0 | 1 | 4 | 0
Not completed — Pregnancy | 1 | 0 | 1 | 0
Not completed — Non-compliance with Study Drug | 1 | 0 | 1 | 0
Not completed — Maximum Clinical Benefit | 2 | 0 | 5 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 2 | 0
Not completed — Participant Request to Discontinue Study Treatment | 4 | 0 | 6 | 0
Not completed — Death | 0 | 2 | 0 | 0
Not completed — Study Drug Toxicity | 1 | 0 | 4 | 0
Not completed — Progressive Disease | 6 | 4 | 7 | 0
Not completed — Not Reported | 0 | 0 | 2 | 0
Not completed — Site Closed | 0 | 1 | 1 | 0
Period: PK Sub-Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | PK Sub-Study
Started | 0 | 0 | 0 | 7 (4 Participants Joined PK Sub-study from Cohort 3)
Completed | 0 | 0 | 0 | 7 (All 7 participants Completed. 4 participants who joined from cohort 3 re-joined Cohort 3 after PK Sub-study completed.)
Not Completed | 0 | 0 | 0 | 0
Period: Follow-Up
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | PK Sub-Study
Started | 21 (Not all participants who discontinued treatment entered the follow-up period) | 12 (Not all participants who discontinued treatment entered the follow-up period) | 47 (Not all participants who discontinued treatment entered the follow-up period) | 0
Completed | 12 | 3 | 25 | 0
Not Completed | 9 | 9 | 22 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 5 | 0
Not completed — Death | 1 | 9 | 0 | 0
Not completed — Lost to Follow-up | 3 | 0 | 0 | 0
Not completed — Reason Not Specified | 4 | 0 | 13 | 0
Not completed — Missing - Administrative Reasons in Russia | 1 | 0 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | PK Sub-Study | Total
Number analyzed (Participants) | 29 | 17 | 84 | 3 | 133
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.60 (4.774) | 12.10 (3.680) | 11.95 (4.418) | 13.33 (1.154) | 12.05 (4.255)
Age, Customized [Number; unit: participants]
  < 2 years | 1 | 0 | 2 | 0 | 3
  >= 2 to < 7 years | 3 | 2 | 10 | 0 | 15
  >= 7 to < 12 years | 6 | 6 | 28 | 0 | 40
  >= 12 to < 18 years | 17 | 9 | 44 | 3 | 73
  >= 18 years | 2 | 0 | 0 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 9 | 39 | 2 | 66
  Male | 13 | 8 | 45 | 1 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 5 | 0 | 7
  Not Hispanic or Latino | 4 | 0 | 20 | 1 | 25
  Unknown or Not Reported | 23 | 17 | 59 | 2 | 101
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 20 | 13 | 56 | 2 | 91
  Black or African American | 2 | 0 | 4 | 0 | 6
  Asian | 6 | 3 | 23 | 0 | 32
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Other | 1 | 1 | 0 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Major Cytogenetic Response (MCyR) Rate
Description: Major Cytogenetic Response (MCyR) rate is defined as the proportion of all treated participants who achieved a complete (0%) or partial (1%-35% Ph+ metaphases in at least 20 metaphases in bone marrow) cytogenetic response, expressed as percentage. The denominator of the MCyR response rate consists of all treated participants in Cohort 1, and the numerator is all participants in Cohort 1 achieving MCyR. 95% confidence interval was calculated by Clopper-Pearson exact method.
Time Frame: From first dose of study therapy until 30 days after last dose (Assessed up to September 2016, approximately 90 months)
Population: Primary efficacy endpoint pre-specified only for participants treated in Cohort 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 29
percentage of participants | 89.7 [72.6 to 97.8]

2. Primary Outcome: Complete Hematologic Response (CHR) Rate
Description: Complete Hematologic Response (CHR) rate is defined as the proportion of all treated participants who achieve a confirmed CHR while on-study, expressed as percentage. CHR is defined as including no more than 5% blasts in bone marrow and normal white blood cell count without blasts in peripheral blood, expressed as percentage. The denominator of the CHR response rate consists of all treated participants in Cohort 2, and the numerator is all participants in Cohort 2 achieving CHR. 95% confidence interval was calculated by Clopper-Pearson exact method.
Time Frame: From first dose of study therapy until 30 days after last dose (Assessed up to September 2016, approximately 90 months)
Population: Primary efficacy endpoint pre-specified only for participants treated in Cohort 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 2
Number analyzed (Participants) | 17
percentage of participants | 29.4 [10.3 to 56.0]

3. Primary Outcome: Complete Cytogenetic Response (CCyR) Rate
Description: Complete Cytogenetic Response (CCyR) rate is defined as the proportion of all treated participants who achieve a CCyR while on-study, expressed as a percentage. CCyR rate is defined as 0% Ph+ metaphases in at least 20 metaphases in bone marrow. The denominator of the CCyR response rate consists of all treated participants in Cohort 3, and the numerator is all participants in Cohort 3 achieving CCyR. 95% confidence interval was calculated by Clopper-Pearson exact method.
Time Frame: From first dose of study therapy until 30 days after last dose (Assessed up to September 2016, approximately 90 months)
Population: Primary efficacy endpoint pre-specified only for participants treated in Cohort 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 3
Number analyzed (Participants) | 84
percentage of participants | 94.0 [86.7 to 98.0]

4. Secondary Outcome: Major Cytogenetic Response (MCyR) Rate in Cohort 2
Description: Major Cytogenetic Response (MCyR) rate was defined as the proportion of all treated participants who achieved a complete (0%) or partial (1%-35% Ph+ metaphases in at least 20 metaphases in bone marrow) cytogenetic response. The percentage of treated participants in each arm with MCyR is reported.
Time Frame: From first dose of study therapy until 30 days after last dose (Assessed up to September 2016, approximately 90 months)
Population: Secondary efficacy endpoint pre-specified only for participants treated in Cohort 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 2
Number analyzed (Participants) | 17
percentage of participants | 52.9 [27.8 to 77.0]

5. Secondary Outcome: Complete Hematologic Response (CHR) Rate in Cohorts 1 and 3
Description: Complete Hematologic Response (CHR) rate defined as the proportion of all treated participants who achieve a confirmed CHR while on-study. CHR is defined as including no more than 5% blasts in bone marrow and normal white blood cell count without blasts in peripheral blood. The percentage of treated participants in each arm with CHR is reported.
Time Frame: From first dose of study therapy until 30 days after last dose (Assessed up to September 2016, approximately 90 months)
Population: Secondary efficacy endpoint pre-specified only for participants treated in Cohort 1 and Cohort 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 | Cohort 3
Number analyzed (Participants) | 29 | 84
percentage of participants | 93.1 [77.2 to 99.2] | 96.4 [89.9 to 99.3]

6. Secondary Outcome: Rate of Best Cytogenetic Response
Description: The number of participants achieving their best on-study cytogenetic response was reported as a percentage of all treated participants in that arm. (Based on >=20 Metaphases)
Time Frame: From first dose of study therapy until 30 days after last dose (Assessed up to September 2016, approximately 90 months)
Population: All treated participants
Measure: Number; unit: percentage of participants
Groups:
- Cohort 3a: Children and adolescents with CP-CML who were treatment-naive received dasatinib tablets at 60 mg/m2 QD on a continuous oral regimen.
- Cohort 3b: Children and adolescents with CP-CML who were treatment-naive received dasatinib powder for oral suspension (PFOS) at 72 mg/m2 QD on a continuous oral regimen.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 3a | Cohort 3b
Number analyzed (Participants) | 29 | 17 | 84 | 51 | 33
percentage of participants
  Complete (0%) | 82.8 | 29.4 | 94.0 | 96.1 | 90.9
  Partial (>0% - 35%) | 6.9 | 23.5 | 2.4 | 2.0 | 3.0
  Minor (>35% - 65%) | 3.4 | 0 | 0 | 0 | 0
  Minimal (>65% - 95%) | 3.4 | 0 | 1.2 | 2.0 | 0
  No Response (>95% - 100%) | 0 | 5.9 | 0 | 0 | 0
  Unable to Determine | 3.4 | 41.2 | 2.4 | 0 | 6.1

7. Secondary Outcome: Time to Major Cytogenetic Response (MCyR)
Description: Time to MCyR is defined as the time from first dose of dasatinib until the first day MCyR criteria are met, computed only for participants whose best response is MCyR. (Based on >=20 Metaphases)
Time Frame: From first dose until MCyR criteria are met (assessed up to September 2016, approximately 90 months)
Population: All treated participants with MCyR
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 3a | Cohort 3b
Number analyzed (Participants) | 26 | 9 | 81 | 50 | 31
months | 3.1 [2.8 to 4.1] | 1.6 [0.5 to 5.7] | 3.0 [2.9 to 4.3] | 3.3 [2.9 to 5.6] | 3.0 [2.8 to 5.0]

8. Secondary Outcome: Duration of Major Cytogenetic Response (MCyR)
Description: Duration of MCyR will be computed from the first day criteria are met for MCyR until the date progressive disease (PD) is reported (or treatment is discontinued for PD) or death. Participants who neither discontinue due to PD nor die will be censored on the date of their last hematologic or cytogenetic assessment, whichever comes last. (Based on >=20 Metaphases)
Time Frame: From first day criteria are met for MCyR until the date PD is reported or death (assessed up to September 2016, approximately 90 months)
Population: All treated participants with MCyR
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 3a | Cohort 3b
Number analyzed (Participants) | 26 | 9 | 81 | 50 | 31
months | NA [54.9 to NA] — Insufficient number of participants with events | 11.2 [0.3 to NA] — Insufficient number of participants with events | NA [52.7 to NA] — Insufficient number of participants with events | NA [52.7 to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events

9. Secondary Outcome: Time to Complete Cytogenetic Response (CCyR)
Description: Time to CCyR is defined as the time from first dose of dasatinib until the first day CCyR criteria are met, computed only for participants whose best response is CCyR. (Based on >=20 Metaphases)
Time Frame: From first dose until CCyR criteria are met, assessed up to September 2016 (approximately 90 months)
Population: All treated participants with CCyR
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 3a | Cohort 3b
Number analyzed (Participants) | 24 | 5 | 79 | 49 | 30
months | 3.9 [2.8 to 5.6] | 1.6 [0.5 to 5.7] | 5.6 [5.0 to 6.0] | 5.7 [3.7 to 6.2] | 5.6 [3.1 to 6.0]

10. Secondary Outcome: Duration of Complete Cytogenetic Response (CCyR)
Description: Duration of CCyR will be computed from the first day criteria are met for CCyR until the date progressive disease (PD) is reported (or treatment is discontinued for PD) or death. Participants who neither discontinue due to PD nor die will be censored on the date of their last hematologic or cytogenetic assessment, whichever comes last. (Based on >=20 Metaphases)
Time Frame: From first day criteria are met for CCyR until the date of progressive disease or death (assessed up to September 2016, approximately 90 months)
Population: All treated participants who achieved CCyR
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 3a | Cohort 3b
Number analyzed (Participants) | 24 | 5 | 79 | 49 | 30
months | NA [54.9 to NA] — Insufficient number of participants with events | NA [1.0 to NA] — Insufficient number of participants with events. | NA [49.9 to NA] — Insufficient number of participants with events | NA [49.9 to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events

11. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as time from the first dosing date until the time PD is first documented by the investigator or death. Participants who die without a reported date of progression will be considered to have progressed on the date of death. Participants who neither progress nor die will be censored on the date of their last cytogenetic or hematologic assessment. Based on Kaplan-Meier methodology. Disease Progression was defined as any of the following criteria: -For CP-CML, progression to AP-CML or BP-CML while at highest tolerated dose -Increasing WBC -Loss of CHR (defined as any of the following: WBC count rises to >20.0x10^9/L; Platelet count rises to >600x10^9/L; appearance of extramedullary disease; appearance of >5% myelocytes+metamyelocytes in blood; appearance of blasts/promyelocytes in peripheral blood) -Loss of MCyR or increase in Ph+ bone marrow cells by >=30% from nadir -Death from any case during treatment.
Time Frame: 174 Months
Population: All treated participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 3a | Cohort 3b
Number analyzed (Participants) | 29 | 17 | 84 | 51 | 33
Months | NA [87.00 to NA] — Insufficient number of participants with events | 6.67 [0.95 to 12.16] | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events

12. Secondary Outcome: Time to Complete Hematologic Response (CHR)
Description: Time to CHR is defined as the time from first dose of dasatinib until the first day CHR criteria are met, provided they are confirmed 4 weeks later, computed only for participants whose best response is CHR.
Time Frame: From first dose until CHR criteria are met, assessed up to September 2016 (approximately 90 months)
Population: All treated participants with CHR
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 3a | Cohort 3b
Number analyzed (Participants) | 27 | 5 | 81 | 51 | 30
months | 0.7 [0.5 to 1.8] | 2.5 [0.5 to 2.8] | 1.2 [0.9 to 1.4] | 1.2 [0.9 to 1.4] | 1.0 [0.7 to 1.8]

13. Secondary Outcome: Duration of Complete Hemotologic Response (CHR)
Description: Duration of CHR will be computed from the first day all criteria are met for CHR, provided they are confirmed 4 weeks later, until the date progressive disease (PD) is reported (or treatment is discontinued for PD) or death. Participants who neither discontinue due to PD nor die will be censored on the date of their last hematologic assessment.
Time Frame: From first day criteria are met for CHR until date of disease progression or death (assessed up to September 2016, approximately 90 months)
Population: All treated participants with CCyR
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 3a | Cohort 3b
Number analyzed (Participants) | 27 | 5 | 81 | 51 | 30
months | NA [NA to NA] — Insufficient number of participants with events | NA [1.9 to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events

14. Secondary Outcome: Disease-Free Survival
Description: Disease free survival is defined as time from CCyR for participants with newly diagnosed chronic phase CML and for participants with chronic phase CML who are resistant or intolerant to imatinib (cohort 3 and cohort 1), and as time from CHR for participants with advanced phase CML and PH + ALL (cohort 2) until the time progression is first documented by the investigator or death from any cause. Based on Kaplan-Meier methodology. (CML: Chronic Myeloid Leukemia).
Time Frame: 168 Months
Population: All treated participants with response of CCyR or CHR
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 3a | Cohort 3b
Number analyzed (Participants) | 24 | 5 | 79 | 49 | 30
Months | NA [75.83 to NA] — Insufficient number of participants with events | NA [1.87 to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events

15. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as time from the first dosing date until the time of death. All participants will be followed yearly for survival for up to 5 years after treatment discontinuation. Participants who have not died or who are lost to follow-up will be censored on the last date the participant is known to be alive. Based on Kaplan-Meier methodology using graphs.
Time Frame: 174 Months
Population: All treated participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 3a | Cohort 3b
Number analyzed (Participants) | 29 | 17 | 84 | 51 | 33
Months | NA [NA to NA] — Insufficient number of participants with events | 13.63 [4.67 to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events

16. Secondary Outcome: Major Molecular Response (MMR) Rate
Description: Molecular response was assessed using BCR-ABL transcript levels measurement by real-time quantitative polymerase chain reaction (qPCR). MMR for participants with the p210 BCR-ABL transcript variant was defined as a ratio BCR-ABL/ABL <= 10-3 or 0.1% on the international scale. In this study, ABL was used as the control-gene. For a participant with the p190 BCR-ABL transcript variant (occurring in Cohort 2 only), on-study assessments were compared to the participant's individual baseline BCR-ABL/ABL ratio and a reduction to < 0.1% or a 3-log reduction from baseline was considered an MMR.
Time Frame: From date of first treatment to date of MMR (assessed up to Jan 2025, approximately 15 years and 10 months)
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 3a | Cohort 3b
Number analyzed (Participants) | 29 | 17 | 84 | 51 | 33
percentage of participants | 69.0 [49.2 to 84.7] | 29.4 [10.3 to 56.0] | 84.5 [75.0 to 91.5] | 90.2 [78.6 to 96.7] | 75.8 [57.7 to 88.9]

17. Secondary Outcome: Complete Molecular Response (CMR) Rate
Description: Molecular response was assessed using BCR-ABL transcript levels measurement by real-time quantitative polymerase chain reaction (qPCR). (CMR) is defined as absence of BCR-ABL rearrangements by real-time qPCR analysis. The percentage of treated participants with CMR is reported by arm.
Time Frame: From date of first treatment to date of CMR (assessed up to Jan 2025, approximately 15 years and 10 months)
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 3a | Cohort 3b
Number analyzed (Participants) | 29 | 17 | 84 | 51 | 33
percentage of participants | 27.6 [12.7 to 47.2] | 11.8 [1.5 to 36.4] | 42.9 [32.1 to 54.1] | 49.0 [34.8 to 63.4] | 33.3 [18.0 to 51.8]

18. Secondary Outcome: Major Cytogenetic Response (MCyR) Rate up to 2 Years
Description: Major Cytogenetic Response (MCyR) rate is defined as the proportion of all treated participants who achieved a complete (0%) or partial (1%-35% Ph+ metaphases in at least 20 metaphases in bone marrow) cytogenetic response. The percentage of treated participants with MCyR is reported by arm.
Time Frame: 24 months
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 3a | Cohort 3b
Number analyzed (Participants) | 29 | 17 | 84 | 51 | 33
percentage of participants
  12 months | 89.7 [72.6 to 97.8] | 58.8 [32.9 to 81.6] | 96.4 [89.9 to 99.3] | 98.0 [89.6 to 100.0] | 93.9 [79.8 to 99.3]
  24 months | 89.7 [72.6 to 97.8] | 58.8 [32.9 to 81.6] | 96.4 [89.9 to 99.3] | 98.0 [89.6 to 100.0] | 93.9 [79.8 to 99.3]

19. Secondary Outcome: Complete Cytogenetic Response (CCyR) Rate up to 2 Years
Description: Complete Cytogenetic Response (CCyR) rate is defined as the proportion of all treated participants who achieve a CCyR while on-study. CCyR rate is defined as 0% Ph+ metaphases in at least 20 metaphases in bone marrow. The percentage of treated participants with CCyR is reported by arm.
Time Frame: 24 months
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 3a | Cohort 3b
Number analyzed (Participants) | 29 | 17 | 84 | 51 | 33
percentage of participants
  12 months | 75.9 [56.5 to 89.7] | 41.2 [18.4 to 67.1] | 92.9 [85.1 to 97.3] | 96.1 [86.5 to 99.5] | 87.9 [71.8 to 96.6]
  24 months | 82.8 [64.2 to 94.2] | 41.2 [18.4 to 67.1] | 94.0 [86.7 to 98.0] | 96.1 [86.5 to 99.5] | 90.9 [75.7 to 98.1]

20. Secondary Outcome: Major Molecular Response (MMR) Rate up to 7.5 Years
Description: Molecular response will be assessed using BCR-ABL transcript levels measurement by real-time qPCR. MMR for participants with the p210 BCR-ABL transcript variant is defined according to the recommendations of Hughes et al. as a ratio BCR-ABL/ABL <= 10-3 or 0.1% on the international scale proposed by the authors. The standardized baseline, as established in the IRIS trial, is taken to represent 100% on the international scale and a 3-log reduction in ratio (BCR-ABL transcripts/ABL or BCR) from the standardized baseline (MMR) is fixed at 0.1%. In this study, ABL or other housekeeping gene, will be used as the control-gene. For a participant with the p190 BCR-ABL transcript variant, on-study assessments will be compared to the participant's individual baseline BCR-ABL/ABL ratio and a reduction to < 0.1% or a 3-log reduction from baseline will be considered an MMR. The percentage of treated participants with MMR is reported by arm.
Time Frame: 90 months
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 3a | Cohort 3b
Number analyzed (Participants) | 29 | 17 | 84 | 51 | 33
percentage of participants
  12 months | 41.4 [23.5 to 61.1] | 29.4 [10.3 to 56.0] | 52.4 [41.2 to 63.4] | 56.9 [42.2 to 70.7] | 45.5 [28.1 to 63.6]
  24 months | 55.2 [35.7 to 73.6] | 29.4 [10.3 to 56.0] | 70.2 [59.3 to 79.7] | 74.5 [60.4 to 85.7] | 63.6 [45.1 to 79.6]
  36 months | 62.1 [42.3 to 79.3] | 29.4 [10.3 to 56.0] | 77.4 [67.0 to 85.8] | 82.4 [69.1 to 91.6] | 69.7 [51.3 to 84.4]
  48 months | 62.1 [42.3 to 79.3] | 29.4 [10.3 to 56.0] | 82.1 [72.3 to 89.6] | 88.2 [76.1 to 95.6] | 72.7 [54.5 to 86.7]
  60 months | 65.5 [45.7 to 82.1] | 29.4 [10.3 to 56.0] | 83.3 [73.6 to 90.6] | 90.2 [78.6 to 96.7] | 72.7 [54.5 to 86.7]
  72 months | 65.5 [45.7 to 82.1] | 29.4 [10.3 to 56.0] | 84.5 [75.0 to 91.5] | 90.2 [78.6 to 96.7] | 75.8 [57.7 to 88.9]
  84 months | 65.5 [45.7 to 82.1] | 29.4 [10.3 to 56.0] | 84.5 [75.0 to 91.5] | 90.2 [78.6 to 96.7] | 75.8 [57.7 to 88.9]
  90 months | 69.0 [49.2 to 84.7] | 29.4 [10.3 to 56.0] | 84.5 [75.0 to 91.5] | 90.2 [78.6 to 96.7] | 75.8 [57.7 to 88.9]

21. Secondary Outcome: Complete Molecular Response (CMR) Rate up to 7.5 Years
Description: Molecular response will be assessed using BCR-ABL transcript levels measurement by real-time quantitative polymerase chain reaction (qPCR). (CMR) is defined as absence of BCR-ABL rearrangements by real-time qPCR analysis. The percentage of treated participants with CMR is reported by arm.
Time Frame: 90 months
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 3a | Cohort 3b
Number analyzed (Participants) | 29 | 17 | 84 | 51 | 33
percentage of participants
  12 months | 6.9 [0.8 to 22.8] | 5.9 [0.1 to 28.7] | 8.3 [3.4 to 16.4] | 9.8 [3.3 to 21.4] | 6.1 [0.7 to 20.2]
  24 months | 17.2 [5.8 to 35.8] | 5.9 [0.1 to 28.7] | 25.0 [16.2 to 35.6] | 33.3 [20.8 to 47.9] | 12.1 [3.4 to 28.2]
  36 months | 17.2 [5.8 to 35.8] | 11.8 [1.5 to 36.4] | 28.6 [19.2 to 39.5] | 33.3 [20.8 to 47.9] | 21.2 [9.0 to 38.9]
  48 months | 24.1 [10.3 to 43.5] | 11.8 [1.5 to 36.4] | 34.5 [24.5 to 45.7] | 43.1 [29.3 to 57.8] | 21.2 [9.0 to 38.9]
  60 months | 24.1 [10.3 to 43.5] | 11.8 [1.5 to 36.4] | 40.5 [29.9 to 51.7] | 47.1 [32.9 to 61.5] | 30.3 [15.6 to 48.7]
  72 months | 24.1 [10.3 to 43.5] | 11.8 [1.5 to 36.4] | 41.7 [31.0 to 52.9] | 49.0 [34.8 to 63.4] | 30.3 [15.6 to 48.7]
  84 months | 24.1 [10.3 to 43.5] | 11.8 [1.5 to 36.4] | 42.9 [32.1 to 54.1] | 49.0 [34.8 to 63.4] | 33.3 [18.0 to 51.8]
  90 months | 27.6 [12.7 to 47.2] | 11.8 [1.5 to 36.4] | 42.9 [32.1 to 54.1] | 49.0 [34.8 to 63.4] | 33.3 [18.0 to 51.8]

ADVERSE EVENTS:
Time Frame: Participants were assessed for All-Cause Mortality, Serious adverse events (SAEs) and Other adverse events (AEs) in all treated participants (up to approximately 14 years 6 months). The participants who crossed over from Cohort 3 to PK Sub-study are accounted for in both arms. PK Sub-study only for the duration of the PK Sub-study.
Groups:
- Cohort 2: BP-CML Only: Children and adolescents with BP-CML who were resistant or intolerant to, or relapsed after imatinib therapy received dasatinib tablets at a dose schedule of 80 mg/m2 QD on a continuous oral regimen.
- Cohort 2: Ph + ALL Only: Children and adolescents with Ph+ ALL who were resistant or intolerant to, or relapsed after imatinib therapy received dasatinib tablets at a dose schedule of 80 mg/m2 QD on a continuous oral regimen.
Arm/Group | Cohort 1 | Cohort 2: BP-CML Only | Cohort 2: Ph + ALL Only | Cohort 3a | Cohort 3b | PK Sub-Study
All-Cause Mortality (participants affected / at risk) | 1/29 | 4/8 | 7/9 | 0/51 | 0/33 | 0/7
Serious Adverse Events (participants affected / at risk) | 16/29 | 7/8 | 6/9 | 21/51 | 12/33 | 0/7
Other Adverse Events (participants affected / at risk) | 27/29 | 7/8 | 9/9 | 50/51 | 33/33 | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=29) | Cohort 2: BP-CML Only (N=8) | Cohort 2: Ph + ALL Only (N=9) | Cohort 3a (N=51) | Cohort 3b (N=33) | PK Sub-Study (N=7)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 3 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 3 | 2 | 2 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 2 | 0 | 0 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 0
Anal ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 1 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 3 | 2 | 0 | 2 | 3 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Adenovirus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 2 | 2 | 0
Device related infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Enterococcal sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 3 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 2 | 0 | 0 | 1 | 2 | 0
Large intestine infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Meningitis aseptic (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Myringitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Upper aerodigestive tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Viral pericarditis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Craniofacial fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Acute lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Blast cell crisis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Chronic myeloid leukaemia transformation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0 | 0 | 0 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 2 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2 | 0 | 0 | 0
Arachnoiditis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Facial nerve disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Personality change (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ischaemic nephropathy (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Genital haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=29) | Cohort 2: BP-CML Only (N=8) | Cohort 2: Ph + ALL Only (N=9) | Cohort 3a (N=51) | Cohort 3b (N=33) | PK Sub-Study (N=7)
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 2 | 11 | 7 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Haemoglobinaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 2 | 0 | 3 | 2 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 6 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 6 | 4 | 3 | 17 | 8 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 4 | 4 | 13 | 8 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 2 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 2 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 2 | 3 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 8 | 3 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 2 | 0 | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 1 | 1 | 0 | 1 | 3 | 0
Eye oedema (Eye disorders) | 0 | 0 | 0 | 1 | 2 | 0
Eye pain (Eye disorders) | 3 | 0 | 2 | 3 | 1 | 0
Periorbital oedema (Eye disorders) | 1 | 0 | 0 | 0 | 2 | 0
Vision blurred (Eye disorders) | 1 | 1 | 0 | 3 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 10 | 1 | 2 | 18 | 12 | 0
Abdominal pain upper (Gastrointestinal disorders) | 7 | 0 | 0 | 12 | 6 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Anal ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 1 | 1 | 3 | 1 | 0
Constipation (Gastrointestinal disorders) | 4 | 2 | 0 | 11 | 5 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0 | 3 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 17 | 3 | 3 | 29 | 16 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 6 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Gingival bleeding (Gastrointestinal disorders) | 2 | 0 | 0 | 2 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 11 | 3 | 2 | 22 | 13 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 2 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 2 | 1 | 3 | 4 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 3 | 0 | 1 | 5 | 1 | 0
Vomiting (Gastrointestinal disorders) | 16 | 3 | 3 | 22 | 13 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 1 | 2 | 0
Chest pain (General disorders) | 2 | 0 | 0 | 2 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 1 | 3 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 3 | 1 | 0
Fatigue (General disorders) | 8 | 1 | 2 | 11 | 8 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 2 | 0
Malaise (General disorders) | 0 | 0 | 1 | 1 | 0 | 0
Mass (General disorders) | 0 | 0 | 0 | 0 | 2 | 0
Mucosal inflammation (General disorders) | 1 | 1 | 0 | 0 | 2 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 3 | 4 | 0
Oedema peripheral (General disorders) | 3 | 1 | 0 | 5 | 3 | 0
Pain (General disorders) | 3 | 1 | 1 | 6 | 6 | 0
Peripheral swelling (General disorders) | 2 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 15 | 1 | 5 | 23 | 14 | 0
Swelling face (General disorders) | 0 | 0 | 0 | 1 | 2 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 2 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 3 | 0
Hypersensitivity (Immune system disorders) | 2 | 0 | 0 | 0 | 1 | 0
Abscess (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 3 | 0 | 0 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 3 | 1 | 0
Conjunctivitis (Infections and infestations) | 4 | 0 | 0 | 2 | 2 | 0
Ear infection (Infections and infestations) | 1 | 0 | 1 | 5 | 5 | 0
Febrile infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 2 | 2 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 1 | 8 | 2 | 0
Gastroenteritis viral (Infections and infestations) | 2 | 0 | 0 | 0 | 1 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 3 | 0 | 0
Gingivitis (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 2 | 0 | 1 | 0 | 1 | 0
Influenza (Infections and infestations) | 3 | 0 | 0 | 9 | 3 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0 | 2 | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
Molluscum contagiosum (Infections and infestations) | 2 | 0 | 0 | 2 | 0 | 0
Nasopharyngitis (Infections and infestations) | 8 | 0 | 0 | 10 | 4 | 0
Oral herpes (Infections and infestations) | 0 | 2 | 0 | 5 | 1 | 0
Otitis media (Infections and infestations) | 1 | 1 | 0 | 1 | 1 | 0
Pharyngitis (Infections and infestations) | 2 | 2 | 2 | 7 | 2 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 2 | 3 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 3 | 0
Rhinitis (Infections and infestations) | 3 | 0 | 1 | 8 | 4 | 0
Sinusitis (Infections and infestations) | 4 | 0 | 1 | 3 | 3 | 0
Skin infection (Infections and infestations) | 2 | 0 | 0 | 1 | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 1 | 0 | 3 | 2 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 3 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 10 | 1 | 1 | 19 | 14 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 3 | 0 | 0
Viral infection (Infections and infestations) | 3 | 0 | 1 | 3 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 3 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 3 | 4 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 2 | 0
Sunburn (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 1 | 1 | 0
Alanine aminotransferase increased (Investigations) | 4 | 3 | 1 | 3 | 6 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 2 | 0 | 4 | 5 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1 | 2 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0 | 3 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0 | 2 | 4 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0
Blood urea increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0 | 0 | 5 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1 | 8 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0 | 2 | 12 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 4 | 1 | 0
Weight increased (Investigations) | 2 | 1 | 0 | 3 | 3 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 2 | 4 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1 | 0 | 4 | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0
Hyperalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 4 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 5 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 2 | 3 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 2 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 1 | 1 | 13 | 9 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 1 | 0 | 12 | 8 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3 | 5 | 0 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 3 | 4 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 2 | 4 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0 | 5 | 6 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 | 2 | 0 | 11 | 15 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 4 | 4 | 0
Arachnoiditis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 1 | 0 | 12 | 3 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Facial paralysis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 17 | 3 | 5 | 25 | 16 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 5 | 0 | 0 | 1 | 1 | 0
Somnolence (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 3 | 1 | 1 | 3 | 3 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 4 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 3 | 4 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 4 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 1 | 1 | 0 | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0 | 4 | 1 | 0
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 2 | 0
Menstruation irregular (Reproductive system and breast disorders) | 2 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 3 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 3 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 1 | 4 | 19 | 12 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 4 | 4 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 5 | 4 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 3 | 3 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 0 | 12 | 11 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 5 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 3 | 4 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 12 | 4 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 2 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3 | 2 | 0
Acne (Skin and subcutaneous tissue disorders) | 4 | 0 | 1 | 2 | 7 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 6 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 2 | 2 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 2 | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 0 | 1 | 2 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1 | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 4 | 3 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 2 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 0 | 0 | 8 | 4 | 0
Rash (Skin and subcutaneous tissue disorders) | 9 | 1 | 1 | 19 | 14 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 3 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 1 | 0 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 4 | 4 | 0
Xeroderma (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 2 | 3 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 5 | 5 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 3 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.